CLINICAL TRIAL: NCT05331924
Title: Quality of Life Improvement in Dry Eye Patients After Intense Pulsed Light Therapy Compared to Punctal Plugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Molham Abdelhafez Elbakary, Assistant professor of Ophthalmology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35345/3/22
Record Dates: First submitted 2022-04-08; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Evaporative Dry Eye
Keywords: Dry eye; MGD; IPL therapy; Punctal plugs
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Punctal Plugs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL therapy (Active Comparator): Fifteen patients with severe to moderate evaporative dry eye disease were treated with 3 sessions of IPL therapy.
  Interventions: Procedure: IPL therapy
- Punctal plugs (Active Comparator): Fifteen patients with severe to moderate evaporative dry eye disease were treated with silicone punctal plug insertion.
  Interventions: Procedure: Punctal plugs

INTERVENTIONS:
Procedure: IPL therapy — Intense pulsed light therapy (IPL) is a non-coherent large wavelength high-intensity light in the range of 500-1200nm. It has been used by many investigators for the treatment of evaporative dry eye safely and effectively.
  Arms: IPL therapy
Procedure: Punctal plugs — Silicone punctal plugs are small pieces of silicone designed to block tear drainage through occluding the lacrimal punctum.
  Arms: Punctal plugs

SUMMARY:
Dry eye disease (DED) is a widely spread disorder of tears and ocular surface affecting hundreds of millions around the world. Manifestations resulting from moderate to severe DED have significant effects on the patient's quality of life (QOL). These patients may suffer pain, role limitation, sleep disorders, anxiety, and depression. QOL affection may be comparable to serious illnesses such as renal failure, angina, and disabling fractures.

Evaporative form is the commonest form of DED and it is mainly caused by meibomian glands dysfunction (MGD). The usual traditional treatment options for MGD include warm compresses, expression of meibomian glands (MG), anti-inflammatory drugs, and lubricant eye drops. In many instances, the traditional treatment with artificial tears is not effective.

Non-pharmacological intervention such as punctal occlusion was advocated in these patients. Punctal plugs are designed to block lacrimal drainage, which helps in the preservation of lubricant drops, improving the tear film quantitively and qualitatively. Intense pulsed light therapy (IPL) is another option that has been used by many investigators for the treatment of evaporative dry eye due to MGD safely and effectively.

This study was conducted to compare the improvement of patients' QOL after treatment of severe to moderate evaporative DED with IPL therapy versus silicone punctal plug insertion.

The study included 30 patients with severe to moderate evaporative dry eye secondary to MGD. The effect of DED on patients' QOL was evaluated with the aid of ocular surface disease index (OSDI) questionnaire. Fifteen patients were treated with IPL therapy. The treatment consisted of 3 sessions, with 15 days between the first and second sessions, and 30 days between the second and third sessions. And 15 patients were treated by silicone punctal plug insertion. After the completion of treatment, the Improvement of patients' QOL was evaluated by OSDI questionnaire. The results of both treatments were compared.

ELIGIBILITY:
Inclusion Criteria:

* MGD patients with moderate to severe evaporative dry eye.
* Patients older than 18 years old.

Exclusion Criteria:

* Patients with dry eye due to auto-immune disorders. e.g.: Sjogren syndrome.
* Patients with conjunctival cicatrizing diseases. e.g.: ocular cicatricial pimphegoid.
* Patients with mild dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Patient's quality of life (QOL) affection. | before treatment
  The effect of dry eye on the patient's Quality Of Life (QOL) was evaluated with the aid of the Ocular Surface Disease Index (OSDI) questionnaire. A score of 33 or more indicated severe affection, 23 to 33 indicated moderate, 13 to 22 mild, while 12 or less represented the normal range.
Change in patient's quality of life (QOL) affection. | Within 1 month after completion of treatment
  The effect of dry eye on the patient's Quality Of Life (QOL) was evaluated with the aid of the Ocular Surface Disease Index (OSDI) questionnaire. A score of 33 or more indicated severe affection, 23 to 33 indicated moderate, 13 to 22 mild, while 12 or less represented the normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided